CLINICAL TRIAL: NCT03006302
Title: Phase 2 Study of Epacadostat, Pembrolizumab, and CRS-207, With or Without Cyclophosphamide and GVAX Pancreas Vaccine in Patients With Metastatic Pancreas Cancer
Brief Title: Epacadostat, Pembrolizumab, and CRS-207, With or Without CY/GVAX Pancreas in Patients With Metastatic Pancreas Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J16173; IRB00118520 (Other: JHMIRB); 5P01CA247886-02 (NIH)
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Results first posted 2024-06-20 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Pancreatic cancer; Vaccine; Immunotherapy; Pembrolizumab; PD-1; IDO; CRS-207; Epacadostat
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — epacadostat; pembrolizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Dose Level 1 (Experimental): Epacadostat/Pembrolizumab/CY/GVAX/CRS-207
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Biological: CRS-207; Drug: Cyclophosphamide; Biological: GVAX Pancreas Vaccine
- Part 1: Dose Level 2 (Experimental): Epacadostat/Pembrolizumab/CY/GVAX/CRS-207
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Biological: CRS-207; Drug: Cyclophosphamide; Biological: GVAX Pancreas Vaccine
- Part 1X: Dose Level 2 (Experimental): Epacadostat/Pembrolizumab/CRS-207
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Biological: CRS-207
- Part 1X: Dose Level 3 (Experimental): Epacadostat/Pembrolizumab/CRS-207
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Biological: CRS-207
- Part 2: Dose Expansion (Experimental): Epacadostat/Pembrolizumab/CRS-207
  Interventions: Drug: Epacadostat; Drug: Pembrolizumab; Biological: CRS-207

INTERVENTIONS:
Drug: Epacadostat — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Epacadostat (100, 300, or 600 mg) is taken by mouth twice a day, every day.
  Other Names: INCB024360
Drug: Pembrolizumab — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on day 1 of Cycles 1-6.
  Other Names: MK-3475; KEYTRUDA
Biological: CRS-207 — CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 10^9 CFU) will be administered IV on Day 2 of Cycles 3-6.
Drug: Cyclophosphamide — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Cyclophosphamide (200 mg/m^2) will be administered IV on day 1 of Cycles 1 and 2.
  Other Names: CY; CYTOXAN
  Arms: Part 1: Dose Level 1; Part 1: Dose Level 2
Biological: GVAX Pancreas Vaccine — Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). GVAX will be administered on Day 2 of Cycles 1 and 2.
  Other Names: GVAX; Panc 10.05 pcDNA-1/GM-Neo, Panc 6.03 pcDNA-1/GM-Neo
  Arms: Part 1: Dose Level 1; Part 1: Dose Level 2

SUMMARY:
This study will enroll patients who have metastatic pancreatic cancer and have progressed on prior chemotherapy.

Part 1 (dose escalation) participants will receive epacadostat/pembrolizumab/cyclophosphamide(CY)/GVAX pancreas vaccine followed by epacadostat/pembrolizumab/CRS-207, Part 1X (dose escalation) participants will receive epacadostat/pembrolizumab/CRS-207. Part 2X (dose expansion) participants will receive epacadostat/pembrolizumab/CRS-207.

The primary objectives of this study are to determine the recommended dose of epacadostat in this combination and assess survival of subjects in both treatment groups.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

* Documented adenocarcinoma of the pancreas
* Have disease progression after prior chemotherapy for metastatic pancreas cancer (or adjuvant or neoadjuvant if progression occurred within 6 months of completing this regimen)
* Presence of at least one measurable lesion
* Patient acceptance to have a tumor biopsy of an accessible lesion at 2 time points (baseline and on study)
* ECOG performance status of 0 or 1
* Life expectancy of greater than 3 months
* Adequate organ and marrow function defined by study-specified laboratory tests

Exclusion Criteria (abbreviated):

* Brain metastases
* Clinical or radiographic ascites (some trace amount may be allowed)
* Rapidly progressing disease
* Live vaccine within 30 days of study treatment (flu vaccine allowed)
* Surgery within 28 days of study treatment (some exceptions for minor procedures)
* Use of an investigational agent or device within 28 days of study treatment.
* Chemotherapy, radiation, or biological cancer therapy within 14 days of study treatment.
* Prior treatment with anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti PD-L2, or with IDO inhibitor.
* Use of growth factors within 14 days of study treatment
* Use of any systemic steroids within 14 days of study treatment or other immunosuppressive agents within 7 days of study treatment.
* Use of more than 2 g/day of acetaminophen
* Use of any UGT1A9 inhibitor
* Use of warfarin
* Use of MAOIs or drugs with significant MAOI activity within the 21 days of screening
* History of Seratonin Syndome
* Known allergy to both penicillin and sulfa
* Known or suspected hypersensitivity to any monoclonal antibody or any study drug component
* Have artificial joints or implants that cannot be easily removed or a history of infection associated with an implant
* Significant or malignant pleural effusion
* New pulmonary embolism, extremity deep venous thromboembolism, or portal vein thrombosis within 2 months of study enrollment
* History of autoimmune disease (exceptions for Graves or Hashimoto's disease, vitiligo, and type I diabetes mellitus)
* Gastrointestinal condition that may affect drug absorption
* Significant heart disease or heart disease requiring antibiotic for prevention of endocarditis
* History of abnormal electrocardiogram (ECG) that is deemed meaningful by the investigator
* History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis
* Pulse oximetry of < 92% on room air or the need for supplemental home oxygen
* Infection with HIV, hepatitis B or hepatitis C
* Other conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access that would affect the patient's ability to comply with study visits and procedures
* Pregnant or breastfeeding women
* Unwillingness or inability to follow the study schedule for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, M.D., Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was excluded from analysis because they did not receive the study drug due to their inability to maintain eligibility after enrollment.
Groups:
- Part 1: Dose Level 1: Epacadostat/Pembrolizumab/CY/GVAX/CRS-207
  Epacadostat: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Epacadostat (100 mg) is taken by mouth twice a day, every day.
  Pembrolizumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on day 1 of Cycles 1-6.
  Cyclophosphamide: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Cyclophosphamide (200 mg/m^2) will be administered IV on day 1 of Cycles 1 and 2.
  GVAX Pancreas Vaccine: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). GVAX will be administered on Day 2 of Cycles 1 and 2.
  CRS-207: CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 10^9 CFU) will be administered IV on Day 2 of Cycles 3-6.
- Part 1: Dose Level 2: Epacadostat/Pembrolizumab/CY/GVAX/CRS-207
  Epacadostat: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Epacadostat (300 mg) is taken by mouth twice a day, every day.
  Pembrolizumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on day 1 of Cycles 1-6.
  Cyclophosphamide: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Cyclophosphamide (200 mg/m^2) will be administered IV on day 1 of Cycles 1 and 2.
  GVAX Pancreas Vaccine: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). GVAX will be administered on Day 2 of Cycles 1 and 2.
  CRS-207: CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 10^9 CFU) will be administered IV on Day 2 of Cycles 3-6.
- Part 1X: Dose Level 2: Epacadostat/Pembrolizumab/CRS-207
  Epacadostat: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Epacadostat (300 mg) is taken by mouth twice a day, every day.
  Pembrolizumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on day 1 of Cycles 1-6.
  CRS-207: CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 10^9 CFU) will be administered IV on Day 2 of Cycles 3-6.
- Part 1X: Dose Level 3; Part 2: Dose Expansion: Epacadostat/Pembrolizumab/CRS-207 Epacadostat: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Epacadostat (600 mg) is taken by mouth twice a day, every day.
  Pembrolizumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on day 1 of Cycles 1-6.
  CRS-207: CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 10^9 CFU) will be administered IV on Day 2 of Cycles 3-6.
Period: Overall Study
Arm/Group | Part 1: Dose Level 1 | Part 1: Dose Level 2 | Part 1X: Dose Level 2 | Part 1X: Dose Level 3 | Part 2: Dose Expansion
Started (Started = enrolled and received at least one dose of study drug) | 6 | 4 | 3 | 7 | 20
Completed (Completed = Received 1 course (6 cycles) of treatment) | 2 | 1 | 2 | 0 | 4
Not Completed | 4 | 3 | 1 | 7 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Dose Level 1 | Part 1: Dose Level 2 | Part 1X: Dose Level 2 | Part 1X: Dose Level 3 | Part 2: Dose Expansion | Total
Number analyzed (Participants) | 6 | 4 | 3 | 7 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 1 | 2 | 12 | 24
  >=65 years | 0 | 1 | 2 | 5 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 1 | 7 | 14
  Male | 5 | 0 | 2 | 6 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 6 | 4 | 3 | 7 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 2 | 3
  White | 5 | 4 | 2 | 7 | 18 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Epacadostat
Description: Dose escalation (part I of the trial only) to determine the maximum tolerated dose (MTD) in mg BID. Epacadostat (100, 300, or 600 mg) was taken by mouth twice a day, every day.
Time Frame: 9 weeks
Population: In Part 1 of the study (Epacadostat dose escalation), six patients were assessed in Dose Level 1 (DL1), seven patients were assessed in Dose Level 2 (DL2), and six patients were assessed in Dose Level 3 (DL3) since one patient was replaced because they came off treatment prior to completing the dose limiting toxicity (DLT) review period.
Measure: Number; unit: mg BID
Groups:
- Part 1: Dose Escalation: Epacadostat/Pembrolizumab/CY/GVAX/CRS-207
  Epacadostat: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Epacadostat (100, 300, or 600 mg) is taken by mouth twice a day, every day.
  Pembrolizumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on day 1 of Cycles 1-6.
  Cyclophosphamide: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Cyclophosphamide (200 mg/m^2) will be administered IV on day 1 of Cycles 1 and 2.
  GVAX Pancreas Vaccine: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). GVAX will be administered on Day 2 of Cycles 1 and 2.
  CRS-207: CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 10^9 CFU) will be administered IV on Day 2 of Cycles 3-6.
Arm/Group | Part 1: Dose Escalation
Number analyzed (Participants) | 19
mg BID | 600

2. Primary Outcome: 6 Month Survival
Description: Number of subjects who are alive 6 months or longer after the date of first treatment.
Time Frame: 6 months
Population: Per the clinical trial design, 6 month survival analyses included all subjects who received the MTD (Dose Level 3). Since the enrollment criteria and dose are the same, combining those who are treated at MTD at both parts increase the power and enable to estimate the treatment effect with increased precision. This included the 6 subjects evaluable in Part 1X portion of the trial and the 20 subjects enrolled in Part 2 portion of the trial for a total of 26 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1X/Part 2: Epacadostat/Pembrolizumab/CRS-207
  Epacadostat: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Epacadostat (600 mg) is taken by mouth twice a day, every day.
  Pembrolizumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on day 1 of Cycles 1-6.
  CRS-207: CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 10^9 CFU) will be administered IV on Day 2 of Cycles 3-6.
Arm/Group | Part 1X/Part 2
Number analyzed (Participants) | 26
Participants | 12

3. Secondary Outcome: Number of Participants Experiencing Drug-Related Adverse Events (AEs) Requiring Treatment Discontinuation
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Level 1 | Part 1: Dose Level 2 | Part 1X: Dose Level 2 | Part 1X: Dose Level 3 | Part 2: Dose Expansion
Number analyzed (Participants) | 6 | 4 | 3 | 7 | 20
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were evaluated for up to 18 months. All-cause mortality was evaluated for up to 67 months. During the survival follow-up portion of the trial, patients were evaluated for all-cause mortality past the time frame for treatment and the assessment of adverse events.
Groups:
- Part 1: Dose Level 1: Epacadostat/Pembrolizumab/CY/GVAX/CRS-207
  Epacadostat: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Epacadostat (100 mg) is taken by mouth twice a day, every day.
  Pembrolizumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on day 1 of Cycles 1-6.
  CRS-207: CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 10^9 CFU) will be administered IV on Day 2 of Cycles 3-6.
  Cyclophosphamide: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Cyclophosphamide (200 mg/m^2) will be administered IV on day 1 of Cycles 1 and 2.
  GVAX Pancreas Vaccine: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). GVAX will be administered on Day 2 of Cycles 1 and 2.
- Part 1: Dose Level 2: Epacadostat/Pembrolizumab/CY/GVAX/CRS-207
  Epacadostat: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Epacadostat (300 mg) is taken by mouth twice a day, every day.
  Pembrolizumab: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Pembrolizumab (200 mg) will be administered IV on day 1 of Cycles 1-6.
  CRS-207: CRS-207: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). CRS-207 (1 × 10^9 CFU) will be administered IV on Day 2 of Cycles 3-6.
  Cyclophosphamide: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). Cyclophosphamide (200 mg/m^2) will be administered IV on day 1 of Cycles 1 and 2.
  GVAX Pancreas Vaccine: Patients will receive treatment every 3 weeks for 6 cycles of treatment within a course (total of 18 weeks). GVAX will be administered on Day 2 of Cycles 1 and 2.
Arm/Group | Part 1: Dose Level 1 | Part 1: Dose Level 2 | Part 1X: Dose Level 2 | Part 1X: Dose Level 3 | Part 2: Dose Expansion
All-Cause Mortality (participants affected / at risk) | 5/6 | 4/4 | 3/3 | 7/7 | 19/20
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/4 | 1/3 | 2/7 | 7/20
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 3/3 | 7/7 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose Level 1 (N=6) | Part 1: Dose Level 2 (N=4) | Part 1X: Dose Level 2 (N=3) | Part 1X: Dose Level 3 (N=7) | Part 2: Dose Expansion (N=20)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Visceral arterial ischemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Volume overload (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IVC stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jejunal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminitis (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Billiary track infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose Level 1 (N=6) | Part 1: Dose Level 2 (N=4) | Part 1X: Dose Level 2 (N=3) | Part 1X: Dose Level 3 (N=7) | Part 2: Dose Expansion (N=20)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (3) | 2 (2) | 0 (0) | 6 (6)
Enlarged lymp nodes (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (7) | 2 (12) | 2 (2) | 5 (13) | 17 (47)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (6) | 4 (8) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudoaneurysm (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear bleading (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (4) | 0 (0) | 3 (3) | 4 (4)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3)
Belching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 3 (3) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Polydipsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic duct stricture (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (10) | 3 (12) | 1 (2) | 2 (3) | 15 (35)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (5) | 0 (0) | 1 (1) | 6 (6)
Chills (General disorders) | 4 (10) | 2 (8) | 3 (13) | 7 (17) | 19 (64)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (5) | 0 (0) | 0 (0) | 2 (2) | 8 (9)
Fever (General disorders) | 3 (5) | 2 (6) | 3 (7) | 5 (16) | 19 (66)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pain at biopsy site (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Groin pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19-infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 2 (4) | 3 (6) | 4 (5) | 11 (14)
Platelet count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (3) | 3 (4) | 2 (2) | 4 (4) | 9 (9)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 8 (26)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (3) | 2 (2) | 7 (17)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cold intolerance-hands and feet (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Depression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 4 (5)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subungual hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 3 (5) | 1 (1) | 2 (2) | 1 (2)
Hypotension (Vascular disorders) | 1 (3) | 2 (10) | 1 (5) | 1 (2) | 8 (13)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
MRSA infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin peeling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccine site erythema (Skin and subcutaneous tissue disorders) | 6 (8) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Vaccine site hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccine site induration (Skin and subcutaneous tissue disorders) | 6 (8) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Vaccine site pain (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Vaccine site pruritis (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
IVC stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03006302/Prot_SAP_000.pdf